CLINICAL TRIAL: NCT06501495
Title: Slow Waves During Sleep and Wakefulness: a Common Denominator for Cognitive and Attentional Disorders in Normal and Pathological Aging (Exploratory Study)
Brief Title: Links Between Cognitive Deficits During Normal or Pathological Aging and Slow Waves Measured in EEG
Acronym: MemoAge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP240231
Record Dates: First submitted 2024-07-01; First posted 2024-07-15 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Aging; Alzheimer Disease
Keywords: aging; Alzheimer's disease; sleep; memory; attention; slow
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- young adults, older adults without cognitive deficits, prodromal Alzheimer's Disease (Experimental): young adults, older adults without cognitive deficits, prodromal Alzheimer's Disease
  Interventions: Other: video polysomnography; Other: Attention task

INTERVENTIONS:
Other: video polysomnography — video polysomnography during 2 nights
Other: Attention task — Attention task : SART Test (Sustained Attention to Response Task)

SUMMARY:
With age, memory processes (encoding, consolidation and retrieval) as well as daytime vigilance are altered. Sleep is also impaired in older adults, notably slow waves that are known to play a key role in memory consolidation. Interestingly, some slow waves can also be detected in EEG recordings during wakefulness, and have been related to vigilance fluctuations.

The investigators believe that slow waves, during both sleep and wakefulness, could constitute a common biomarker of sleep disturbances and daytime vigilance problems. A dysregulation of slow waves could thus explain the impact of aging on the different memory processes. Since alterations in memory capacity, attention, and sleep quality are further exacerbated in patients with Alzheimer's disease (AD), the investigators propose to study the links between aging (normal and pathological), sleep and daytime vigilance alterations, and their impacts on the different key stages of memory.

The investigators will examine the associations between slow waves and changes in memory and vigilance in normal and pathological aging by studying young adults, seniors without cognitive disorders, and patients with prodromal AD. By replaying sensory cues associated with learning material during sleep, the investigators will also evaluate the effectiveness of auditory stimulation during sleep to enhance memory consolidation in older adults without and without cognitive deficits.

Overall, this study aims to better understand the relationships between slow waves, aging, memory, and vigilance, providing insights into cognitive decline and potential interventions in aging and Alzheimer's disease.

DETAILED DESCRIPTION:
Introduction Aging is accompanied by cognitive decline, particularly affecting memory functions. Additionally, both the quantity and quality of sleep decrease with advancing age, specifically altering sleep oscillations (such as slow waves) that are involved in the reactivation of memories and are thus central to memory consolidation.

Aging is also associated with difficulties in maintaining daytime vigilance, even after a period of rest, impacting cognitive function, including the encoding and retrieval of memories. Interestingly, recent studies have revealed the existence of sleep intrusions, in the form of slow waves, in wakefulness EEG recordings. These have been associated with subjective and objective markers of fatigue, predict transient lapses in attention, and are particularly present after sleep deprivation. the investigators believe that slow waves, during both sleep and wakefulness, could constitute a common biomarker of sleep disturbances and daytime vigilance problems. A dysregulation of slow waves (fewer during sleep, more during wakefulness) could thus explain the impact of aging on the three fundamental stages of the memory process (encoding, consolidation, and retrieval). Since alterations in memory capacity, attention, and sleep quality are further exacerbated in patients with Alzheimer's disease (AD), the investigators propose to study the links between aging (normal and pathological), sleep and daytime vigilance alterations, and their impacts on the different key stages of memory.

Aims Our main objective is to test the associations between slow waves (during sleep and wakefulness) and the alterations in memory and vigilance during normal and pathological aging by studying young adults, seniors without cognitive disorders, and patients of the same age with prodromal AD.

Additionally, the investigators aim to test the efficiency of targeted memory reactivation (TMR) in older adults with and without cognitive deficits. TMR is a technique that has been showed to boost memory consolidation in young adults and mice by replaying during sleep sensory cues that have been previously associated with the learning material.

Methods Participants To do so, the stydy will include three groups: young adults (18-35 y.o), older adults without cognitive deficits (65-80 y.o), and older adults of the same age and with cognitive deficits (patients with prodromal Alzheimer's disease). Prodromal stage of Alzheimer's disease diagnosis will be performed by trained neurologists at the at the Memory and Alzheimer's Disease Institute (IM2A) of the Pitié-Salpêtrière Hospital, according to international diagnostic criteria as a clinical phenotype of progressive amnestic syndrome of the hippocampal type, associated with biological markers of Alzheimer's disease from lumbar puncture (Aβ < 600 pg/mL and ptau > 60 pg/mL). During their clinical follow-up at the IM2A, patients diagnosed with prodromal AD will be offered the opportunity to participate in the study, in agreement with their attending physician. Healthy volunteers (both young and elderly) will be recruited through public announcements via the Relay for Information on Cognitive Sciences (RISC), from patients' relatives, or through the Fondation Recherche Alzheimer. Participation of both patients and healthy individuals will be voluntary, free, and informed. Participants will be contacted (by phone or email) by one of the study investigators. They will be informed about the conduct and purpose of the research protocol.

Protocol All participants will spend 3 days in the Sleep Disorders Unit of the Salpêtrière Hospital, including two nights.

Day 1: Participants will arrive in the late afternoon and will be fitted with the sensors required for video-polysomnography to monitor vigilance and sleep stages throughout the experiment. Then, they will 1) complete an attention task (modified version of the Sustained Attention to Response Task, SART), 2) perform an associated memory task (old/new task) consisting on recognition of words they have seen in the SART task, and 3) their resting-state EEG activity will be recorded. They will sleep in the laboratory (night 1, without intervention).

Day 2: Participants will retake the word recognition task the morning after night 1. During the afternoon they will fill different sleep questionnaires to assess their subjective feeling about their sleep: Pittsburgh sleep quality index (PSQI), Epworth sleepiness scale and the REM Behavior Disorder Screening Questionnaire (RBDSQ), as well as the geriatric depression scale (GDS). In the late afternoon, they will perform the learning and test phases of the visuospatial memory task. They will then sleep in the laboratory (night 2, with TMR). During their slow-wave sleep, half of the sounds associated with the items from the visuospatial memory task will be replayed.

Day 3: Participants will once again perform the visuospatial memory test the morning after night 2.

ELIGIBILITY:
* Common Inclusion Criteria for All Three Groups:

Male or female Signed informed consent Affiliated with a social security system Native French speakers Completed at least 7 years of schooling (minimum 9th grade level)

Specific Inclusion Criteria for Each Group:

Patients:

Age: 60 to 85 years Prodromal stage of Alzheimer's disease diagnosed according to international diagnostic criteria, characterized by a clinical phenotype of progressive amnesic syndrome of the hippocampal type, associated with biological markers of Alzheimer's disease from lumbar puncture (Aβ < 600 pg/mL and ptau > 60 pg/mL)

Cognitively Healthy Seniors:

Age: 60 to 85 years Age and sex matched with the Patients group "Cognitively healthy" status defined by a score of ≥ 26 on the MMSE (Mini-Mental State Examination), a score of ≥ 16 on the BREF (Batterie Rapide d'Efficience Frontale), and a score of ≥ 8 on the 5-word test

Young Adults:

Age: 18 to 35 years Sex matched with the Patients group "Cognitively healthy" status defined by a score of ≥ 26 on the MMSE (Mini-Mental State Examination), a score of ≥ 16 on the BREF (Batterie Rapide d'Efficience Frontale), and a score of ≥ 8 on the 5-word test

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
slow waves density | 2 days
  quantifying slow waves with their density (during sleep, wakefulness at rest and during tasks)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Teichmann, MD, Principal Investigator — assisitance publique Hôpitaux de paris
Locations (1):
- Maladies du Sommeil, Paris, France

REFERENCES:
- See also: Project article on the funder's website (Fondation France Alzheimer) — https://alzheimer-recherche.org/16423/regulation-locale-du-sommeil-vieillissement-et-fonctions-cognitives/